CLINICAL TRIAL: NCT00120237
Title: A Placebo-Controlled Randomized Trial of Misoprostol in the Management of the Third Stage of Labor in the Home Delivery Setting in Rural Pakistan
Brief Title: Misoprostol for the Prevention of Postpartum Hemorrhage in Rural Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Aga Khan University (Other); Aga Khan Health Services (Other); The Aga Khan Foundation (Other); Family Care International (Other)
Responsible Party: Gynuity Health Projects, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2.4.4
Record Dates: First submitted 2005-07-07; First posted 2005-07-15 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Postpartum Hemorrhage; Anemia
Keywords: Postpartum hemorrhage; Misoprostol; Maternal morbidity; Developing countries; Traditional birth attendants
MeSH Terms: conditions — Postpartum Hemorrhage; Anemia | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Misoprostol — 600 mcg oral misoprostol administered during third stage of labor

SUMMARY:
This community-based trial will study misoprostol for the prevention of postpartum hemorrhage in rural Pakistan. Traditional birth attendants assisting home deliveries will administer study tablets (600 mcg oral misoprostol or placebo) in the third stage of labor to women participating in the trial. Blood loss, hemoglobin levels, side effects, and other variables will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in general good health, home delivery
* Must live in one of 78 study villages

Exclusion Criteria:

* Hypertension
* Non-cephalic presentation
* Polyhydramnios
* Previous cesarean section
* Suspected multiple pregnancy
* Suspected still birth
* Antepartum hemorrhage
* Previous complication in 3rd trimester
* Anemia of <8 g/dl

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Postpartum hemorrhage (blood loss >or= 500 mL) | Measured at 1 hour postpartum or until active bleeding has stopped
Drop in hemoglobin > 2 g/dL from pre to post-delivery | Hemoblobin (Hb) level measured 3-5 days after delivery

SECONDARY OUTCOMES:
Intermediate and severe PPH (blood loss >or=750 mL and >or= than 1000 mL) | Blood loss measured at 1 hr postpartum or until active bleeding stopped
Mean blood loss | blood loss measured at 1 hr postpartum or until active bleeding stopped
Side effects experienced among recently delivered mothers | Interviews conducted 1 day post-delivery
Anemia (<9 g/dL and <11 g/dL) | Postpartum hemoglobin assessed 3 days post-delivery

CONTACTS AND LOCATIONS:
Overall Officials: Gijs Walraven, MD, Principal Investigator — Aga Khan Health Services; Juanita Hatcher, PhD, Principal Investigator — Aga Khan University; Naushaba Mobeen, MD, Study Director — Aga Khan University; Jennifer Blum, MPH, Study Director — Gynuity Health Projects; Zafar Ahmad, MD, Study Director — Aga Khan Health Services; Nadeem Zuberi, MD, Study Director — Aga Khan University; Jill Durocher, Study Director — Gynuity Health Projects
Locations (1):
- Home delivery setting, Chitral, Chitral District, Pakistan

REFERENCES:
- See also: Gynuity Health Projects — http://www.gynuity.org